CLINICAL TRIAL: NCT02845570
Title: Evaluation of Somatostatin Receptor Imaging Using PET/MRI as a Novel Approach to Detecting Pathology in Pulmonary TB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DOTANOC TB
Record Dates: First submitted 2016-07-17; First posted 2016-07-27 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2016-07

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga-DOTANOC PET/MRI (Experimental): Comparison between 68Ga-DOTANOC PET/MRI and 18F-FDG PET/MRI scans
  Interventions: Other: 68Ga-DOTANOC PET/MRI; Other: 18F-FDG PET/MRI

INTERVENTIONS:
Other: 68Ga-DOTANOC PET/MRI
Other: 18F-FDG PET/MRI

SUMMARY:
Imaging using 68Ga-DOTANOC PET (positron emission tomography) has the potential to detect granulomas in pulmonary tuberculosis, leading to previously unexplored indications for this PET tracer, including identification of subclinical disease in latently infected individuals. This study aims to assess the ability of 68Ga-DOTANOC PET/MRI to detect pulmonary lesions in individuals with active pulmonary tuberculosis.

DETAILED DESCRIPTION:
Granulomas, the hallmark of tuberculosis (TB) infection, have an increased density of somatostatin receptors. Somatostatin analog PET tracers, such as 68Ga-DOTANOC, may be able to identify these pulmonary granulomas. Although currently used for other medical indications, 68Ga-DOTANOC PET scanning has not previously been used to detect TB lesions.

This is a pilot study which aims to assess the ability of 68Ga-DOTANOC PET/MRI to detect pulmonary lesions in individuals with active pulmonary tuberculosis. The 68Ga-DOTANOC PET scan and 'standard' 18F-fludeoxyglucose (FDG) PET scan will be compared to enable analysis of differences in uptake between these tracers in terms of number, size and distribution of lesions.

Demonstrating the clinical utility of 68Ga-DOTANOC in active pulmonary TB is necessary prior to using this PET tracer to further explore other potential uses in TB such as identifying individuals with latent TB who are at risk of progressing to active TB, measuring therapeutic response to TB treatment and identifying extrapulmonary lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years and above
2. Willing to comply with the study visits and procedures
3. Willing and able to provide written informed consent
4. Clinical diagnosis of pulmonary TB with characteristic symptoms and compatible X-ray findings plus microbiological confirmation with one or more of (i) Acid fast bacilli (AFB) smear-positive or (ii) molecular test positive or (iii) TB culture positive
5. Not on TB treatment or have completed less than 28 days of TB treatment

Exclusion Criteria:

1. Diabetes that is, in the judgment of the investigator, so poorly controlled that it would prevent adequate PET scanning
2. Cardiac pacemaker, aneurysm clip or other metallic implant considered unsafe for MRI
3. Known chronic kidney disease
4. Occupation involving substantial exposure to radiation
5. Malignancy requiring chemotherapy or radiation
6. Women who are currently pregnant or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value (SUV) of 68Ga-DOTANOC in pulmonary TB lesions using PET/MRI | Within 28 days of commencing TB treatment

SECONDARY OUTCOMES:
Comparison of uptake of 68Ga-DOTANOC with that of 18F-FDG in pulmonary TB. | Within 28 days of commencing TB treatment
  Different uptake values between and within the pulmonary lesions will be measured and compared between the 2 tracers.
Establishment of optimal timing for a 68Ga-DOTANOC PET scan to evaluate TB lung pathology | Over 90 minutes from injection of tracer
  The net tracer uptake rate for 68Ga-DOTANOC (Ki) will be derived from kinetic analysis in combination with dynamic imaging and the relationship between SUV and Ki.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore